CLINICAL TRIAL: NCT03640585
Title: The Effects of Music Therapy on Gross Motor Functions, Pain and Level of Functional Independence in Children With Cerebral Palsy
Brief Title: Effects of Music Therapy in Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, TOMRIS DUYMAZ, Asst. Prof. Ph.D., Istanbul Bilgi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBU2015
Record Dates: First submitted 2018-08-18; First posted 2018-08-21 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Music therapy; Gross motor function
MeSH Terms: conditions — Cerebral Palsy | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: The patients were randomized and divided into 2 groups of 20 people. A randomized list is prepared in a computer environment by a statistician for randomization. In this list, the odd numbers for the control group and the MT group were given double numbers. The group identification is printed on sequentially numbered cards placed in sealed envelopes. After enrollment, the numbered envelope was opened by the patient and the blind investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music therapy (Experimental): Children listened to Classical music disc for 45 minutes.Children treated by neurodevelopmental therapy while listening to this music.A total of 15 treatments were administered for 5 weeks, 3 sessions per week for all patients.
  Interventions: Other: Music therapy
- Control (Placebo Comparator): Only the neurodevelopmental therapy was applied in the control group without music. A total of 15 treatments were administered for 5 weeks, 3 sessions per week for all patients. The sessions were 45 minutes.
  Interventions: Other: Music therapy

INTERVENTIONS:
Other: Music therapy — Only the neurodevelopmental therapy was applied in the second group without music. A total of 15 treatments were administered for 5 weeks, 3 sessions per week for all patients. The sessions were 45 minutes.
  Other Names: Control

SUMMARY:
Purpose:To observe the effects of music therapy on gross motor functions, pain and functional independence measurement in children with cerebral palsy(CP).

Methods:Forty children with CP between 5-11years of age,were randomly divided into a music therapy(MT)+Neurodevelopmental techniques(NDT)group and only NDT group.Children listened to Classical music disc for 45 minutes.Children treated by NDT while listening to this music.Children were evaluated with Gross Motor Function Measurement(GMFM-88),WeeFIM for functional independence measurement,Wong-Baker faces pain rating scale (FACES) for pain intensity before,at the end of treatment and after 3 months of treatment.The treatments were given 3 times in every week,and totally 15 treatments were applied for 5 weeks.

DETAILED DESCRIPTION:
Participants Forty children with spastic CP between the ages of 5 and 11 years were enrolled in this study. Children were classified according to the Gross Motor Function Classification System. The patients were randomized and divided into 2 groups of 20 people. A randomized list is prepared in a computer environment by a statistician for randomization. In this list, the odd numbers for the control group and the MT group were given double numbers. The group identification is printed on sequentially numbered cards placed in sealed envelopes. After enrollment, the numbered envelope was opened by the patient and the blind investigator. The researcher started the session by placing the proper disc CD player before the beginning of the work. Children from 5 to 11 years of age, who had a spastic type CP diagnosis and were able to understand the commands as co-operative, with no hearing problems between GMFCS levels I and III were included in the study. Acute and chronic infectious diseases, coagulation diseases, progressive cerebral diseases such as neoplasms, inherited diseases such as trisomy 21 syndrome, hearing loss, surgery from the upper and lower extremity in the last 1 year, psychiatric problems, weak cooperatives were excluded from the study.

Study design Neurodevelopmental therapy was applied in the first group music accompaniment and only the neurodevelopmental therapy was applied in the second group without music. A total of 15 treatments were administered for 5 weeks, 3 sessions per week for all patients. The sessions were 45 minutes. Classical music is preferred as a musical style. The exercises performed in the musical accompaniment are made according to the rhythms in the music. The treatment schedule is planned so that the commands given to the illness and the movements required to be removed are made in the presence of rhythms. The age and body mass index (BMI) of all patients were recorded. Children were evaluated with Gross Motor Function Measurement (GMFM-88), WeeFIM for functional independence measurement, Wong-Baker faces pain rating scale (FACES) for pain intensity before, at the end of treatment and after 3 months of treatment. Outcome measures are described in more detail below. According to the power analysis results, when the number of enough participants was reached, the study was stopped. Ethics committee approval for the study was obtained from the Istanbul Science University Ethics Committee for Clinical Researches.

ELIGIBILITY:
Inclusion Criteria:

* Children from 5 to 11 years of age
* Who had a spastic type CP diagnosis
* able to understand the commands as co-operative
* no hearing problems
* between GMFCS levels I and III

Exclusion Criteria:

* Acute and chronic infectious diseases
* Coagulation diseases
* Progressive cerebral diseases such as neoplasms
* Inherited diseases such as trisomy 21 syndrome
* Hearing loss
* Surgery from the upper and lower extremity in the last 1 year
* Psychiatric problems
* Weak cooperatives

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-12-03 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-09-23 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measurement | 15 minutes
  The gross motor functions of children with CP have been evaluated with the Gross Motor Function Measurement (GMFM-88), which has been widely used in recent years. There are 5 main divisions. It consists of a total of 88 items consisting of 17 in the supine, prone position and turning section, 20 in the sitting section, 14 in the crawling-laptops section, 13 in the standing section and 24 in the walking-running-stair climbing section. Score 0- The movement can not start. 1- Actively initiates a certain amount of movement (<10%) 2- Completely completes the movement but can not finish (10% - 90%). 3- Completes the movement independently. Each section score is calculated within itself as a percentage, then the five percent score is summed, divided by 5, and the total percentile score is found

SECONDARY OUTCOMES:
Functional independence measurement (WeeFIM) | 5 minutes
  It is a useful, short, comprehensive method of measuring functional, educational, and socially functional limitations of children with CP and other developmental disabilities. The WeeFIM includes 6 items in total, 18 items including self care, sphincter control, transfers, locomotion, communication, social and cognitive. In performing the functions of each item in these areas, the score is scored from 1 to 7, depending on whether or not they get help, whether they do it on time, or whether an auxiliary device is needed. When the task is done with help completely 1; 7 is considered to be totally independent, at the appropriate time and in a safe manner. 1-7 points are awarded depending on the amount of the help. Accordingly, scores of at least 18 (fully dependent) and 126 (fully independent) can be taken
Pain of extremities | 1 minute
  FACES is a pain severity scale that scales from 0 to 10, which can be determined by the child's face expressions without the need for communication that will force them to express the pain they feel when they are 3 years old and older. 0 points means no pain at all, 10 points means severe pain at irresistible levels

CONTACTS AND LOCATIONS:
Overall Officials: TOMRIS DUYMAZ, Principal Investigator — Istanbul Bilgi University
Locations (1):
- Tomris Duymaz, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided